CLINICAL TRIAL: NCT00999635
Title: A Comparison of Functional and Prefabricated Insoles Used for the Preventative Management of Neuropathic Diabetic Foot Ulceration: a Single Blind Randomised Control Trial
Brief Title: A Comparison of Insoles Used to Prevent Neuropathic Diabetic Foot Ulceration
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Plymouth (Other)
Collaborators: Cornwall and Illes of Scilly Primary Care Trust (Unknown); Plymouth Teaching Primary Care Trust (Unknown); Diabetes UK (Other)
Responsible Party: Dr Joanne Paton, University of Plymouth
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 05/Q2103/150
Record Dates: First submitted 2009-10-21; First posted 2009-10-22 (Estimated); Last update posted 2009-10-27 (Estimated); Status verified 2009-10

CONDITIONS: Diabetes; Neuropathic Foot
Keywords: Insoles; Prevention of Ulceration; Diabetic Foot; Neuropathic
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Foot | interventions — Foot Orthoses

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Custom made insole (Experimental): Custom made functional moulded insole
  Interventions: Device: Insole
- Prefabricated Insole (Active Comparator): Prefabricated accommodative moulded insole
  Interventions: Device: Insole

INTERVENTIONS:
Device: Insole — Comparison of custom made and prefabricated insoles designed for the neuropathic diabetic foot, issued for day time wear and followed for a 6 month period

SUMMARY:
Importance of the topic:

Lower extremity amputation is a costly complication of diabetes for both the NHS and the patient. Amputation may be avoided if the preceding foot ulceration can be prevented. One method of reducing the risk of ulceration in the neuropathic foot is through the provision of therapeutic insoles. The type of insole prescribed (prefabricated verses custom made) is currently based on anecdotal evidence. The idea held by many practitioners that the custom made insole is superior in its effect remains speculation, unsupported by the evidence. In the absence of economic analysis, the available data suggests that the custom insole is substantially more expensive to the NHS. This study, to determine which of two types of insole used in therapeutic shoes reduces peak pressure more in the at-risk diabetic foot, is therefore a very important topic and will provide both useful evidence for the NHS podiatry services. It is of course also very important for patients with diabetes as the personal suffering of those undergoing amputation is immense.

The study is a single blind randomised controlled trial comparing custom made with 'off the shelf' insoles.

DETAILED DESCRIPTION:
Aim The study compared custom-made functional insoles with prefabricated insoles for the preventative management of neuropathic diabetic feet, assessing effects on peak pressure, forefoot pressure time integral, total contact area, forefoot rate of loading, duration of load as a percentage of stance, quality of life, perceived foot health and cost.

Method Pilot work investigating the physical properties of materials used to fabricate insoles informed material selection. A single-blind randomised control trial recruited 119 neuropathic participants with diabetes from two Primary Care Trusts and randomly allocated them to either custom-made functional insoles or prefabricated insoles. Data was collected at issue and 6-month follow-up, using the F-scan in-shoe pressure measurement system. Patient perceptions were assessed with the Bristol Foot Score and Audit of Diabetes Dependant Quality of Life. Further analyses were carried out on two subgroups; 1) insole effect on peak pressure in 44 participants with pronated feet, over a 6-month follow-up period; 2) insole durability, investigated in a second subgroup of 60 participants for 12-months. Durability was evaluated in terms of change in insole thickness and reduction in peak pressure.

To increase the robustness of results, data analysis was calculated using three strategies; 1) pure intention-to-treat analysis, including all 119 participants randomised to an intervention; 2) intention-to-treat analysis, using all available data; 3) as-treated analysis, including those participants self-reporting full insole compliance, defined as 60% or more daytime wear.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed as having Type 1 or 2 diabetes mellitus, (recorded within the case notes and confirmed by participant),
* diagnosed with diabetic peripheral neuropathy
* palpable or biphasic pulses
* intact from lower limb vascular or neuropathic ulceration, scoring Grade 0 on the Wagner classification for foot ulcer
* able to walk a minimum of 10 metres unaided
* willing to comply with the requirements of the study.

Exclusion Criteria:

* presented with current or recently healed ulceration less than 6 months prior to study enrolment,
* severe fixed mid-foot or rearfoot deformity e.g. charcot joint, unsuitable for prefabricated insoles and non- bespoke footwear,
* history of major bone or joint surgery of the lower limb including major amputation
* unable to comprehend simple instructions and comply with the study protocols and procedures.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2006-03; Primary Completion 2007-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Reduction in peak pressure | 6-months

SECONDARY OUTCOMES:
Comparison of cost | 6-months

CONTACTS AND LOCATIONS:
Overall Officials: Ray Jones, Professor, Study Director — University of Plymouth; Joanne Paton, PhD, Principal Investigator — University of Plymouth
Locations (2):
- United Kingdom (2):
  - Liskeard Community Hospital, Liskeard, Cornwall
  - Local Care Center Mount Gould, Plymouth, Devon

REFERENCES:
- [Derived] Paton JS, Stenhouse EA, Bruce G, Zahra D, Jones RB. A comparison of customised and prefabricated insoles to reduce risk factors for neuropathic diabetic foot ulceration: a participant-blinded randomised controlled trial. J Foot Ankle Res. 2012 Dec 5;5(1):31. doi: 10.1186/1757-1146-5-31. PMID 23216959